CLINICAL TRIAL: NCT05697107
Title: A Large Scale, Multicenter, Real-World Study on Patients With Advanced GIST Receiving Ripretinib
Brief Title: Ripretinib in Chinese Patients With Advanced GIST: a Real World Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Sun Yat-sen University (Other); Fudan University (Other); Xiangya Hospital of Central South University (Other); Fujian Medical University Union Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); First Affiliated Hospital of Chongqing Medical University (Other); RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shen Lin, Director of GI oncology Affiliation: Peking University, Peking University, Peking University
Other Study IDs: GIST-R-RWD-001
Record Dates: First submitted 2023-01-15; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Ripretinib Oral Tablet — Oral kinase inhibitor

SUMMARY:
to evaluate the clinical efficacy, safety and predictive factors of ripetinib in Chinese patients with advanced GIST in the real world

DETAILED DESCRIPTION:
Ripretinib has become the standard ≥ 4L treatment in advanced GIST. Given the small sample size of patients in the China bridging study of INVICTUS as well as the short marketing time of ripretinib, further exploration on the long-term efficacy and safety of ripretinib, as well as the dominant gene mutation type of ripretinib in Chinese GIST patients is required. Hence, we plan to further explore the efficacy of ripretinib, predictors of efficacy, etc. by collecting and analyzing real-world data from Chinese patients with advanced GIST recieving ripretinib.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years old

* Histologically confirmed gastrointestinal stromal tumor (GIST)
* At least one measurable lesion (mRECIST v1.1)
* Received or receiving ripretinib treatment

Exclusion Criteria:

* Patients who received <1 cycle of ripretinib treatment
* Medical records are incomplete

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed gastrointestinal stromal tumor
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | approximately 7 months
  To assess the efficacy (progression-free survival [PFS]

SECONDARY OUTCOMES:
DCR | approximately 6 months
  To assess disease control rate (DCR)
OS | approximately 12 months
  to assess median overall survival (mOS)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
UNDECIDED

REFERENCES:
- [Derived] Zhang X, Zhang P, Qiu H, Fang Y, Liu H, Zhou Y, Xu H, Yu J, Zhang J, Wang M, Shen L, Li J. Large-Scale, Multicenter, Prospective Registry Study of Ripretinib in Advanced GIST: A Real-World Study from China. Adv Ther. 2023 Sep;40(9):3817-3829. doi: 10.1007/s12325-023-02576-0. Epub 2023 Jun 25. PMID 37356078